CLINICAL TRIAL: NCT02808663
Title: Assessment of the Predictive Value of Fecal Calprotectin for the Outcome of Severe Alcoholic Hepatitis
Acronym: CALPRO-HAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PA14069
Record Dates: First submitted 2016-06-15; First posted 2016-06-22 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Severe Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Blood Specimen Collection

ARMS (1):
- Severe Alcoholic Hepatitis (Experimental)
  Interventions: Biological: fecal calprotectin concentration; Biological: blood collection

INTERVENTIONS:
Biological: fecal calprotectin concentration
Biological: blood collection

SUMMARY:
Severe alcoholic hepatitis, defined by a "Maddrey discriminant function" above 32, is associated with significant short-term mortality. In patients with liver disease, studies have shown alterations of intestinal bacterial flora and an increase in intestinal permeability leading to bacterial translocation across the intestinal barrier. The mechanism involved may be an activation of intestinal macrophages with a local release of cytokines like interleukin-8 (IL-8).

Calprotectin is a protein present in large amounts in the cytosol of neutrophils. Its presence in feces is related to neutrophil migration in intestinal lumen. Thus, fecal calprotectin may be used as a marker of intestinal inflammation. There is evidence that fecal calprotectin levels are increased in cirrhotic patients dependent on the severity of the disease. The predictive value of fecal calprotectin for the outcome of severe alcoholic hepatitis has never been evaluated.

The main objective of this study was to determine if the initial level of fecal calprotectin and its variation after 7 days had a predictive value for the outcome of severe alcoholic hepatitis. Secondary objectives were to determine if fecal calprotectin concentration was correlated with blood concentration of Lipopolysaccharide (LPS) binding protein and predictive of infections.

DETAILED DESCRIPTION:
Severe alcoholic hepatitis, defined by a "Maddrey discriminant function" above 32, is associated with significant short-term mortality. In patients with liver disease, studies have shown alterations of intestinal bacterial flora and an increase in intestinal permeability leading to bacterial translocation across the intestinal barrier. The mechanism involved may be an activation of intestinal macrophages with a local release of cytokines like IL-8.

Calprotectin is a protein present in large amounts in the cytosol of neutrophils. Its presence in feces is related to neutrophil migration in intestinal lumen. Thus, fecal calprotectin may be used as a marker of intestinal inflammation. There is evidence that fecal calprotectin levels are increased in cirrhotic patients dependent on the severity of the disease. The predictive value of fecal calprotectin for the outcome of severe alcoholic hepatitis has never been evaluated.

The main objective of this study was to determine if the initial level of fecal calprotectin and its variation after 7 days had a predictive value for the outcome of severe alcoholic hepatitis. Secondary objectives were to determine if fecal calprotectin concentration was correlated with blood concentration of LPS binding protein and predictive of infections.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe alcoholic hepatitis defined by a "Maddrey discriminant function" above 32
* histological confirmation of the diagnosis and indication for corticotherapy
* signed written informed consent and social security affiliation

Exclusion Criteria:

* age below 18
* pregnant or breastfeeding women
* history of intestinal disease, digestive haemorrhage
* treatment with antibiotics, NSAIDs or proton pump inhibitors during the month before inclusion
* patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-05-06; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
fecal calprotectin concentration | Day1
fecal calprotectin concentration | Day7

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France